CLINICAL TRIAL: NCT00772343
Title: A Phase II Randomized, Placebo-Controlled, Double-Blind, Dose Ranging Study of A Clostridium Difficile Toxoid Vaccine (ACAM-CDIFF™) in Subjects With Clostridium Difficile Infection (CDI)
Brief Title: Study of a Clostridium Difficile Toxoid Vaccine (ACAM-CDIFF™) in Subjects With Clostridium Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: H-030-011; 2008-004907-69 (EudraCT Number); 28439/0001/001 (Other: MHRA)
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Diarrhea; Clostridium Difficile Infection
Keywords: Diarrhea; Clostridium difficile infection; Clostridium difficile toxoid
MeSH Terms: conditions — Diarrhea; Clostridium Infections | interventions — Saline Solution; Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Vaccine (Placebo Comparator): 0.9% Normal saline
  Interventions: Biological: 0.9% Normal Saline
- Low dose (Experimental): Low dose vaccine with adjuvant
  Interventions: Biological: Clostridium difficile toxoid vaccine
- High dose 1 (Experimental): High-dose vaccine with adjuvant
  Interventions: Biological: Clostridium difficile toxoid vaccine with adjuvant
- High dose 2 (Experimental): High-dose vaccine without adjuvant
  Interventions: Biological: Clostridium difficile toxoid vaccine

INTERVENTIONS:
Biological: 0.9% Normal Saline — 0.5 mL, intramuscular on Days 0, 7, and 28
  Other Names: Normal Saline
  Arms: Placebo Vaccine
Biological: Clostridium difficile toxoid vaccine — 0.5 mL, intramuscular on Days 0, 7, and 28
  Other Names: ACAM-CDIFF™
  Arms: Low dose
Biological: Clostridium difficile toxoid vaccine with adjuvant — 0.5 mL, intramuscular on Days 0, 7, and 28
  Other Names: ACAM-CDIFF™; ACAM-CDIFF™ Adjuvant
  Arms: High dose 1
Biological: Clostridium difficile toxoid vaccine — 0.5 mL, intramuscular on Days 0, 7, and 28
  Other Names: ACAM-CDIFF™
  Arms: High dose 2

SUMMARY:
Primary objective: To compare the event rate of CDI in groups assigned to ACAM-CDIFF™ vaccine versus placebo in the 9 week period after the third dose of the study vaccine in subjects with first episode of CDI receiving antibiotics standard of care.

Secondary objective: To evaluate the safety of all dose groups of ACAM-CDIFF™ vaccine versus placebo in subjects with first episode of CDI receiving antibiotics standard of care.

DETAILED DESCRIPTION:
This study is designed primarily to obtain information on the preliminary efficacy, safety and immunogenicity of ACAM-CDIFF™ vaccine, as compared to placebo in subjects who are experiencing their first event of CDI and are being treated with the antibiotic standard of care. This study will be conducted in the United States and United Kingdom. Adult subjects with limited chronic disease, who are currently receiving treatment for their first episode of CDI will be enrolled in this trial. Subjects will be required to be able to take oral antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects, 18 - 85 years old, who understand the risks and benefits of participation and have provided written informed consent for the study.
2. Subjects who are experiencing a first event of CDI diagnosed within the last 10 days.
3. Subjects who are medically stable.
4. Subjects who are willing and able to comply with the study procedures and visit schedules outlined.

Exclusion Criteria:

1. Subjects who are currently on treatment for a recurrence of CDI.
2. Subjects who are currently or have recently been treated with immunoglobulin therapy.
3. Pregnant or breast feeding females.
4. Concurrent, acutely life-threatening diseases.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Recurrence of Clostridium difficile infection. | Approximately 13 weeks after last injection

SECONDARY OUTCOMES:
Safety and immunogenicity | Approximately 13 weeks after last injection.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (31):
- United States (5):
  - Tampa, Florida
  - Marietta, Georgia
  - Worcester, Massachusetts
  - Butte, Montana
  - Rapid City, South Dakota
- United Kingdom (26):
  - Birmingham Heartlands Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Bradford Royal Infirmary, Bradford
  - Royal Sussex County Hospital, Brighton
  - Southmead Hospital, Bristol
  - Frenchay Hospital, Bristol
  - St Helier Hospital, Carshalton
  - Cheltenham Royal Hosptial, Cheltenham
  - St. Richard's Hospital, Chichester
  - New University Hospital (Walsgrave site), Coventry
  - Ninewells Hospital, Dundee
  - West Park Hospital, Epsom
  - Gloucestersh Royal Hospital, Gloucester
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Whittington Hospital, London
  - North Manchester General Hospital, Manchester
  - Royal Oldham Hospital, Manchester
  - St Mary's Hospital, Portsmouth
  - Queen Alexandra Hospital, Portsmouth
  - Northern General Hospital, Sheffield
  - Royal Hallamshire Hospital, Sheffield
  - Stepping Hill Hospital, Stockport
  - Sunderland Royal Hospital, Sunderland
  - St. George's Hospital, Tooting, London
  - Worthing General Hospital, Worthing

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com